CLINICAL TRIAL: NCT04169152
Title: Cap-assisted Endoscopic Sclerotherapy for Internal Hemorrhoids and Rectal Prolapse: a National Multi-centre Prospective Cohort Study
Brief Title: CAES for Internal Hemorrhoids and Rectal Prolapse
Status: Recruiting | Type: Observational
Sponsor: Faming Zhang (Other)
Responsible Party: Sponsor-Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Organization: The Second Hospital of Nanjing Medical University (Other)
Other Study IDs: CAES-CN-191111
Record Dates: First submitted 2019-11-13; First posted 2019-11-19 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Internal Hemorrhoid; Rectal Prolapse
Keywords: Cap-assisted endoscopic sclerotherapy; Internal Hemorrhoid; Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Internal hemorrhoids and rectal prolapse: Participants were treated with Cap-assisted endoscopic sclerotherapy (CAES).
  Interventions: Procedure: Cap-assisted endoscopic sclerotherapy

INTERVENTIONS:
Procedure: Cap-assisted endoscopic sclerotherapy — Cap-assisted endoscopic sclerotherapy (CAES) is an innovation technique for having advantages in accurately controlling the injection angle, direction, depth under direct vision of flexible endoscope.

SUMMARY:
Cap-assisted endoscopic sclerotherapy (CAES) is a new interventional therapy for internal hemorrhoids and rectal prolapse under colonoscopy. However, the long-term efficacy and safety of CAES in the treatment of internal hemorrhoids and rectal prolapse are still not clear due to the lack of large sample studies. Therefore, a nationwide multi-center, large sample, prospective and cohort study was designed to evaluate the efficacy and safety of CAES in the treatment of internal hemorrhoids and rectal prolapse, to provide reliable evidence for popularization of this minimally invasive technology.

DETAILED DESCRIPTION:
CAES is an innovative endoscopic sclerotherapy procedure which is different from traditional method. Firstly, the cap added to the front of colonoscope can fully expose the operating field. Secondly, before or during the opportunity of CAES, endoscopist can perform endoscopic differentiation diagnosis (such as tumors, inflammatory bowel disease and others induced hematochezia), endoscopic therapy within lower-gut based on the same colon preparation, thus saving patients' medical cost, physical and mental pain. The last but not least, specially designed length of endoscopic injection needle (eg.10-20 mm) was used in CAES could be helpful for accurately controlling the injection angle, direction, depth under direct vision and to avoid iatrogenic injury due to ectopic injection.The core value of CAES for internal hemorrhoids and rectal prolapse is to provide precise therapy, reduce the iatrogenic injuries, avoid pain during and after therapy. Our pilot studies demonstrated that CAES based on long injection needle is an effective, safe, convenient operation technique. 100% of participants underwent CAES showed sustained clinical efficacy within the 3-month follow-up, with no severe or obvious complications related to CAES. However, the long-term efficacy and safety of CAES in the treatment of internal hemorrhoids and rectal prolapse need to be confirmed by further large sample real world studies.

ELIGIBILITY:
Inclusion Criteria:

1. Grade I-III internal hemorrhoids (with or without external hemorrhoids) or/and recal prolapse.
2. Patients with bowel preparation.

Exclusion Criteria:

1. History of anoscopic/endoscopic sclerotherapy.
2. Acute thrombotic hemorrhoids or grade IV internal hemorrhoids.
3. Anal stenosis, perianal and perirectal abscess, anal fissure, fistula, fecal incontinence and other severe complications (such as severe anal pain).
4. Inflammatory bowel disease.
5. Full-thickness rectal prolapse through the anus.
6. Acute diarrhea in the past 24 hours.
7. Hypertensive with uncontrolled blood pressure.
8. Cerebrovascular accident.
9. Blood coagulation dysfunction.
10. Pregnant women.
11. Mental disorders.
12. Decompensated cirrhosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Grade I-III internal hemorrhoids and/or rectal prolapse
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 1st week to 24th week
  Recurrence rate defined as the proportion of patients with recurrent hemorrhoids at 24 weeks post-CAES, as derived from patients' self-reported answer. Patients will be considered to have recurrent hemorrhoids when any of the following are recorded: (1) "Unchanged or worse compared with before starting treatment" at 24th week as reported by the patient, or (2) seeking repeat CAES treatment, alternative non-surgical/surgical treatments for internal hemorrhoids within 24weeks (except medication treatment), or (3) presence of any symptoms or events that strongly indicated recurrent hemorrhoids among patients not meeting (1) or (2).

SECONDARY OUTCOMES:
Improvement rate | 1st day, 1st week, 2nd week and 24th week
  Bleeding, prolapse, and anal pain had resolved or remitted after CAES. Bleeding is divided into three degrees: 1. No bleeding; 2. 2: occasionally; 3: quite often.There are three degrees of prolapse: 1. No prolapse; 2: occasionally; 3: quite often.NRS pain digital rating scale was adopted, that is, 0-10 was used to represent different degrees of pain, 0 was painless, and 10 was severe pain. 0 painless, 1-3 mild pain (pain does not affect sleep), 4-6 moderate pain, 7-9 severe pain (inability to fall asleep or waking up during sleep), 10 severe pain.
Failure rate | 1st day, 1st week, 2nd week and 24th week
  Bleeding, prolapse, and anal pain remained the same after CAES. Bleeding is divided into three degrees: 1. No bleeding; 2. 2: occasionally; 3: quite often.There are three degrees of prolapse: 1. No prolapse; 2: occasionally; 3: quite often.NRS pain digital rating scale was adopted, that is, 0-10 was used to represent different degrees of pain, 0 was painless, and 10 was severe pain. 0 painless, 1-3 mild pain (pain does not affect sleep), 4-6 moderate pain, 7-9 severe pain (inability to fall asleep or waking up during sleep), 10 severe pain.
Three-level EuroQol five dimensions (ED-5Q) health scale scores | 24th week
  The ED-5Q questionnaire includes five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), with three levels in each dimension (no/moderate/severe problem). Through the Chinese time trade-off (TTO) value table, the health status of five dimensions will be converted into a preference weight of a ED-5Q index score for further analysis.
Adverse events (AEs) | 1st day, 1st week, 2nd week and 24th week
  AEs refer to adverse medical events that occurs during or after CAES, including bleeding, anal pain, having difficulties in passing gas and defecation, infection, ulcer/bleeding in the injection points under endoscopic examination (5-7 days after CAES) and other symptoms.
severe adverse events (SAEs) severe adverse events (SAEs) severe adverse events (SAEs) Severe adverse events (SAEs) | 1st day, 1st week, 2nd week and 24th week
  SAEs include serious complications directly or indirectly related to the CAES, such as death, bleeding, perforation, infection.
Participants' attitudes toward CAES | 24th week
  The survey on the satisfaction with CAES efficacy, and the willingness to recommend CAES to others.
Symptom severity score | 1day and 24 weeks
  Symptom severity score: five questions about hemorrhoidal symptoms (anal pain, prolapse, itching, soiling, and blood loss) will be self-assessed by patients by answering how often each symptom was encountered (never, sometimes, weekly, or daily). The score is the sum of the points from all five questions, ranging from 0 to 15 points, where an increase in number is an increase in symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD,PhD, Study Chair — The Second Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang T, Xu LJ, Xiang J, He Z, Peng ZY, Huang GM, Ji GZ, Zhang FM. Cap-assisted endoscopic sclerotherapy for hemorrhoids: Methods, feasibility and efficacy. World J Gastrointest Endosc. 2015 Dec 25;7(19):1334-40. doi: 10.4253/wjge.v7.i19.1334. PMID 26722615
- [Background] Tomiki Y, Ono S, Aoki J, Takahashi R, Sakamoto K. Endoscopic sclerotherapy with aluminum potassium sulfate and tannic acid for internal hemorrhoids. Endoscopy. 2014;46 Suppl 1 UCTN:E114. doi: 10.1055/s-0034-1364884. Epub 2014 Mar 27. No abstract available. PMID 24676816
- [Background] Tokunaga Y. Clinical utility of sclerotherapy with a new agent for treatment of rectal prolapse in patients with risks. J Clin Gastroenterol. 2014 Apr;48(4):356-9. doi: 10.1097/MCG.0b013e318299cab8. PMID 23751842